CLINICAL TRIAL: NCT06848218
Title: Music Therapy During NIV Implantation in Pediatric Intensive Care Units
Acronym: MusiNIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RECHMPL23_0191
Record Dates: First submitted 2025-01-23; First posted 2025-02-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Failure (ARF); Non Invasive Ventilation (NIV)
Keywords: Music Therapy; Non invasive Ventilation; Pediatric intensive care unit; Pain; Comfort
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized controlled study, with blinded assessment of primary endpoint.
Who Masked: Outcomes Assessor
Masking Description: the primary endpoint (FLACC Score) will be assessed on patient videos taken during NIV initiation. Thus, 2 FLACC score assessors will be blinded to the randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non invasive ventilation setting with Music Therapy (Experimental): Each child will benefit non invasive ventilation setting for acute respiratory distress.
  In this group, it will be with Music Therapy. Every time, the preparation will be the same with equipment installation with headphones for music listening, in order to keep comparability and blind for the evaluation. Sound will be activated in this group.
  Each child will be videotaped during the non invasive ventilation setting.
  Interventions: Other: Music Therapy; Procedure: Setting Up NIV
- Non invasive ventilation setting without Music Therapy (Sham Comparator): Each child will benefit Non invasive ventilation setting for acute respiratory distress.
  In this group, it will be without Music therapy. Every time, the preparation will be the same with equipment installation with headphones for music listening, in order to keep comparability and blind for the evaluation. Sound will not be activated in this group.
  Each child will be videotaped during the non invasive ventilation setting.
  Interventions: Procedure: Setting Up NIV

INTERVENTIONS:
Other: Music Therapy — This procedure is carried out using headphones installed in the child's ears. The music will be activated if the child is in the Music group, and will not be activated but present if the child is not in the Music group.
  NIV implementation will begin after 10 min of listening. The listening period will continue until the nadir period (when the music is slowest, for maximum relaxation), until 10 min after the start of the NIV.
  Arms: Non invasive ventilation setting with Music Therapy
Procedure: Setting Up NIV — Non invasive ventilation is set up in several stages, with the help of at least two caregivers. The patient will be placed in a half-seated position or seated. Installation begins with the placement of the non invasive ventilation mask harness around the child's head, followed by the application of the mask to the face, held by a caregiver. Once the mask has been applied, ventilation is started by connecting the non invasive ventilation circuit to the mask. The harness is then tightened by the second caregiver.

SUMMARY:
Non-invasive ventilation makes it possible to avoid intubation and improve patients' quality of life. However, pain is associated with discomfort and could lead to failure of this technique.

The aim of this study is to measure the effectiveness of music therapy on pain levels during non-invasive ventilation in critically ill children.

To this end, a pain score (Face Legs Activity Cry Consolability FLACC) will be assessed by raters blinded to the randomization arm during NIV initiation.

The FLACC score will be compared before and during implementation of NIV between two groups: a control group (without music therapy) and an experimental group (with music therapy).

DETAILED DESCRIPTION:
Patient admitted to a Pediatric Intensive Care Unit are exposed to moderate to severe pain due to disease severity and invasive treatment or procedures.

Non invasive ventilation is an essential support in the treatment of infants and children with acute respiratory failure. Acceptance and tolerance are the keys to its success.

Comfort management, including pain management, is most often achieved through the administration of analgesic and/or sedative drugs (analgesics, anti-inflammatories, anxiolytics, hypnotics). However, these therapies, although effective, are not without risks, including potentially serious adverse effects (excessive sedation, prolonged hospitalization and ventilation, tolerance phenomena, withdrawal syndrome, delirium, constipation, etc.). These undesirable effects and their deleterious consequences prompt a more comprehensive approach to patient management, optimizing therapeutic strategies with the common aim of improving patient comfort and pain relief. One specific program, "Music Care" is based on a "U sequence" which use tempo and rhythm variations following the U scheme, to relax patients.

This program will be evaluated in the pediatric intensive care department and the investigators will study the effects on the pain level during a non invasive ventilation setting for children with respiratory failure.

the investigators will compare the variation of the FLACC scores (before and during nopn invasive ventilation setting) to show a difference between both methods. The order (with or without) will be randomized.

ELIGIBILITY:
Target population : Children aged 0 to 17, hospitalized in the pediatric intensive care unit for respiratory failure with indication for NIV.

Inclusion Criteria:

* Children aged 0 to 17 inclusive
* Children hospitalized in pediatric intensive care unit
* Indication for NIV

Exclusion Criteria:

* - Severe deafness
* Clinical condition requiring immediate initiation of NIV
* Refusal to allow the child to be photographed
* Child not assessable by FLACC score (paralysis of lower limbs, etc.)
* Child already receiving NIV respiratory support at home
* Participation in other ongoing research involving the human person at major risk and constraint (RIPH category 1) or a drug trial according to European regulation 536/2014.
* Absence of affiliation to a French social security scheme or beneficiary of such a scheme.
* Subject deprived of liberty (art.L. 1121-6 du CSP)
* Failure to obtain free and informed written or oral consent and authorization to take photographs from both parents (or from a single parent if the patient is accompanied by only one parent, in accordance with article 1122-2 of the French Public Health Code) or from the legal guardian and/or child.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain variation before and during non invasive ventilation setting with and without music therapy. | assessment for 10 minutes before NIV start-up and for 10 minutes during NIV installation
  FLACC (Face Legs Activity Cry Consolability) : The main assessment tool is a simple, rapid behavioral pain assessment scale, commonly used in the pediatric intensive care unit.
  For each item, 3 possible scores: 0 or 1 or 2; the total score is from 0 (no pain) to 10 (severe pain).
  The primary outcome is variation of the Face Legs Activity Cry Consolability (FLACC) score (range, 0-10) comparing before and during non invasive ventilation setting.
  The first FLACC score evaluation will be just before the beginning of music. The Second FLACC score evaluation will be during the non invasive ventilation setting.
  FLACC score evaluation over a 10-minute period, with selection of the highest score for each item during the evaluation period FLACC scores' evaluation will be done from videotape records without by 2 investigators The FLACC score will be determined blindly by two assessors who did not participate in the care, using the video taken when the NIV was set up.

SECONDARY OUTCOMES:
Pain variation during and after non invasive ventilation setting with and without music therapy. the highest score for each parameter will be selected for each evaluation period of 10 minutes | assessment for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  FLACC (Face Legs Activity Cry Consolability) : The main assessment tool is a simple, rapid behavioral pain assessment scale, commonly used in the pediatric intensive care unit.
  For each item, 3 possible scores: 0 or 1 or 2; the total score is from 0 (no pain) to 10 (severe pain).
  The primary outcome is variation of the Face Legs Activity Cry Consolability (FLACC) score (range, 0-10) comparing before and during non invasive ventilation setting.
  The first FLACC score evaluation will be just before the beginning of music. The Second FLACC score evaluation will be during the non invasive ventilation setting.
  FLACC scores' evaluation will be done from videotape records without by 2 investigators
  The FLACC score will be determined blindly by two assessors who did not participate in the care, using the video taken when the NIV was set up.
Physiological data variations between the 2 groups: HR | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  HR: heart rate in beats per minute the highest score for each parameter will be selected for each evaluation period of 10 minutes
Physiological data variations between the 2 groups: FR | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  FR: respiratory rate in inhalations per minute the highest score for each parameter will be selected for each evaluation period of 10 minutes
Physiological data variations between the 2 groups: SBP | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  SBP: systolic blood pressure in millimeters of mercury mmHg the highest score for each parameter will be selected for each evaluation period of 10 minutes
Physiological data variations between the 2 groups: MAP | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  MAP: mean arterial pressure in millimetres of mercury mmHg the highest score for each parameter will be selected for each evaluation period of 10 minutes
Physiological data variations between the 2 groups: SpO2 | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  SpO² : blood oxygen saturation in percent the highest score for each parameter will be selected for each evaluation period of 10 minutes
Physiological data variations between the 2 groups: FiO2. | assessment for 10 minutes before NIV start-up, for 10 minutes during NIV installation and for 10 minutes after NIV start-up
  An initial reading will be taken 10 minutes before NIV start-up, during start-up and 10 minutes afterwards.
  FiO2: fraction of inspired oxygen in percent the highest score for each parameter will be selected for each evaluation period of 10 minutes
NIV set-up time between groups | from initiation to completion of NIV installation
  time from initiation to completion of NIV installation in minutes
Total NIV duration between groups | From initiation of the first NIV to the date of death or discharge from hospital, or up to 1 month after initiation of the NIV at the most
  in hours
Failure to implement NIV between groups | From initiation of the first NIV to the date of death or discharge from hospital, or up to 1 month after initiation of the NIV at the most
  in raw numbers
Use of sedative or anxiolytic drugs during NIV implantation between groups | from initiation to completion of NIV installation
  dose in μg/kg/h
Length of stay in intensive care between groups | from the date of admission in intensive care until discharge, or up to 1 month after initiation of NIV
  in days
total length of hospital stay between groups | from the date of admission to hospital until discharge, or up to 1 month after initiation of NIV
  in days
comparison of the number of NIV-related complications between the 2 groups | from the date of admission to hospital until discharge, or up to 1 month after initiation of NIV
  Number of Complications of NIV, e.g. pneumothorax, decreased cardiac output (hypotension), gastric and abdominal distension, inhalation, nose, face and scalp pressure points, non-compliance, eye irritation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de MONTPELLIER, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided